CLINICAL TRIAL: NCT04463680
Title: The Effect of Rifampin on Etonogestrel Concentrations in Contraceptive Implant Users
Brief Title: Rifampin and the Contraceptive Implant
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 19-2829
Record Dates: First submitted 2020-07-06; First posted 2020-07-09 (Actual); Results first posted 2023-05-09 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Contraception; Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Will receive 2 week regimen of rifampin 600mg per day
  Interventions: Drug: Rifampin 600 MG

INTERVENTIONS:
Drug: Rifampin 600 MG — Administered daily for 2 weeks

SUMMARY:
It is important for women taking rifampin to be aware if they are at greater risk of an unintended pregnancy while on the implant. An unintended pregnancy has many social, emotional, and financial impacts on women and society. Rifampin is also a Class C medication for pregnancy and could have potential negative effects on a developing fetus. Additionally, women considering rifampin for treatment of LTBI face additional risks with an unintended pregnancy, making the reliability of contraception even more important for these women. The results of this study can directly inform counseling on a national and international basis for women who use the contraceptive implant and are considering their treatment options for LTBI.

DETAILED DESCRIPTION:
Rifampin is an antibiotic historically prescribed as part of a treatment regimen for active tuberculosis (TB) infection. Though active TB infections have become rarer over time in the US, it is estimated that up to 13 million people in the US may have latent TB infections (LTBIs), with even greater numbers of LTBIs worldwide1. In efforts to combat the persistent rate of LTBI, the US Centers for Disease Control and Prevention (CDC) released updated treatment guidelines for LTBI in 20181. This recommended treatment guideline consists of four treatment regimens, varying in duration from 3 to 9 months. The CDC recommends utilization of the shorter regimens when possible to achieve higher patient compliance and infection clear rates. The second shortest duration treatment regimen (4 months) consists of daily rifampin only1.

In addition to its antitubercular properties, rifampin is a known strong cytochrome P-450 (CYP) 3A4 enzyme inducer2. Similar to other strong CYP3A4 enzyme inducers (e.g. carbamazepine), rifampin can affect the serum concentrations of exogenous steroid hormones found in hormonal contraception2. The only published literature on the interaction between rifampin and hormonal contraception has focused on combined oral contraceptives3. Five studies that investigated the pharmacokinetics of combined oral contraceptives all found significant reductions in serum ethinyl estradiol and progestin concentrations with rifampin co-administration3. This pharmacokinetic effect is significant enough to warrant a category 3 recommendation (theoretical or proven risks usually outweigh the advantages) from the CDC Medical Eligibility Criteria (MEC) for Contraceptive Use for concomitant rifampin and combined hormonal contraceptive methods4. This pharmacokinetic effect is large enough to raise concerns for combined hormonal contraceptive method efficacy and recommendation of alternative methods. One of those alternative methods is the etonogestrel (ENG) implant (Nexplanon®), which has a category 2 recommendation in the CDC MEC for concomitant rifampin use4. However, in the clarifications for this recommendation, the CDC MEC warns that rifampin is "likely to reduce the effectiveness" of the ENG implant, with no supporting evidence provided4.

Prior work found that a strong CYP3A4 inducer (carbamazepine) caused clinically significant reductions in serum etonogestrel concentrations among contraceptive implant users5. The investigators found a median decrease in serum ENG of 61% (range 25-87) with 8/10 participants having serum ENG concentrations <90pg/mL after concomitant carbamazepine5. Though there is currently no published data on the pharmacokinetic interaction between rifampin and the ENG implant, given its similar enzyme induction properties, there is concern that the CDC MEC recommendation for rifampin and the ENG implant may underestimate the potential risk for contraceptive failure.

Given the social, financial, and healthcare costs of unintended pregnancies, it is imperative that the investigators better understand the drug-drug interaction between rifampin and the ENG implant. Especially in light of the contradictory category 2 recommendation and clarification in the CDC MEC4, more data are needed to determine if rifampin has a significant enough pharmacokinetic effect on the ENG implant to potentially cause contraceptive failure. This information would allow healthcare providers around the world the ability to provide improved counseling to patients needing treatment for LTBI in regards to both their TB treatment regimen and their concurrent contraceptive options.

Specific Aim:

* To evaluate the pharmacokinetic effect of rifampin on serum etonogestrel concentrations in contraceptive implant users at the dose of rifampin used for latent tuberculosis infection (LTBI) treatment (600mg per day)
* Exploratory Aim - to evaluate the effect of rifampin on serologic measures of ovulatory suppression (estradiol and progesterone) in contraceptive implant users

Hypothesis:

· The investigators hypothesize that rifampin will have a significant pharmacokinetic effect on participants' etonogestrel levels resulting in etonogestrel concentrations at least 35% decreased from baseline measurements.

Methods:

The investigators propose a prospective, pre and post study to evaluate the pharmacokinetic effect of rifampin on serum ENG levels in contraceptive implant users. The investigators will enroll healthy women using an ENG implant for at least 12 months and no greater than 36 months.

Participants will then begin a 2 week regimen of rifampin at 600mg per day. This dose is the recommended dose for treatment of LTBI and duration of 2 weeks will achieve steady state rifampin levels with adequate time for liver enzyme induction. All participants will then return at the end of the second week for a repeat blood draw. The investigators will again obtain serum as described above for planned measurement of serum ENG concentrations. The investigators will also obtain blood samples for repeat measurements of serum estradiol and progesterone. The investigators will also measure a serum rifampin level at the time of the second ENG blood draw to confirm compliance. Serum estradiol, serum progesterone, and serum rifampin levels will all be measured at the UCH Clinical Laboratory. At the conclusion of enrollment, all stored serum samples will be de-identified and shipped to a Merck® laboratory for serum ENG concentration measurement. Batch analysis will be performed using a liquid chromatography mass-spectrometry method that has been previously validated. Participants will serve as their own controls for this study.

All participants will be required to use either a back-up non-hormonal method of birth control or abstain from intercourse during the study and for 2 weeks after the last dose of rifampin. Rifampin has a half-life of 3-4 hours, and thus, will be eliminated within 1-2 days of the last dose, but the investigators will allow a full 2 weeks of buffer to ensure that the contraceptive effect of the implant has reinitiated before recommending resuming unprotected intercourse.

All study visits will occur at the Comprehensive Women's Health Clinic in Lowry.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women, who have had an ENG implant for 12-36 months at the time of enrollment and will maintain their implant during the study without modifications.

Exclusion Criteria:

* o Women who are taking any known cytochrome P-450 3A4 enzyme inducers or inhibitors.

  * Women with a known allergy or insensitivity to rifampin.
  * Women with a body mass index (BMI) <18.5, as underweight women may have altered metabolism. The investigators will not have an upper BMI cut-off as studies have shown that overweight and obese women have equivalent metabolism and efficacy with the ENG contraceptive implant6,7.

    • Exclusions Criteria (screening laboratory testing)
  * Women with any hepatic or renal dysfunction as determined by a comprehensive metabolic panel. For purposes of this study, liver function tests will be evaluated and evidence of hepatic dysfunction will be defined as an ALT >52 or AST >39, which are beyond the reference range of normal values used by the University of Colorado clinical laboratory. Renal function will be assessed by a serum creatinine and a value >1.2 will be evidence of renal dysfunction as this is greater than the reference range used by the University of Colorado clinical laboratory.
  * Women with any abnormal hematology as determined by a complete blood count. For purposes of this study, abnormal hematology will be defined as a WBC, RBC, or PLT value beyond the reference range of normal values used by the University of Colorado clinical laboratory.
  * Women with abnormal coagulation factors as determined by coagulation factor tests (PT/INR, PTT). For purposes of this study, abnormal coagulation factors will be defined as any test value beyond the reference range of normal values used by the University of Colorado clinical laboratory.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-02-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Rifampin 600 mg: Will receive 2 week regimen of rifampin 600mg per day
  Rifampin 600 MG: Administered daily for 2 weeks
Period: Overall Study
Arm/Group | Rifampin 600 mg
Started | 24
Completed | 15
Not Completed | 9
Not completed — Not eligible due to laboratory criteria | 5
Not completed — Not eligible due to implant duration of use | 1
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Rifampin 600 mg
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: years] | 28.2 [21.8 to 34.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15
Body mass index [Median (Full Range); unit: kg/m^2] | 25.2 [18.9 to 37.3]
Duration of implant use [Median (Full Range); unit: months] | 22 [12 to 32]

OUTCOME MEASURES:

1. Primary Outcome: Serum Etonogestrel Concentrations
Description: Blood drawn before and after rifampin administration (2 weeks) for serum extraction and etonogestrel analysis
Time Frame: 2 weeks
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Rifampin 600 mg
Number analyzed (Participants) | 15
pg/mL
  Baseline | 164.0 [94.4 to 265.0]
  Post-rifampin | 47.8 [24.7 to 82.8]

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Rifampin 600 mg
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-08): https://cdn.clinicaltrials.gov/large-docs/80/NCT04463680/Prot_SAP_000.pdf